CLINICAL TRIAL: NCT02395965
Title: Use and Effectiveness of Osteopathic Manipulative Medicine (OMM) in the Clinical Setting
Brief Title: OMM Utilization in the Clinical Setting
Status: Completed | Type: Observational
Sponsor: A.T. Still University of Health Sciences (Other)
Collaborators: American Osteopathic Association (Other)
Responsible Party: Sponsor
Other Study IDs: OMM Utilization AOA 11-04-634
Record Dates: First submitted 2015-02-19; First posted 2015-03-24 (Estimated); Last update posted 2015-03-24 (Estimated); Status verified 2014-01

CONDITIONS: Conditions Treated With OMT
Keywords: Osteopathic manipulative medicine; Osteopathic manipulative treatment

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The SPECIFIC AIM of this research study is to evaluate the utilization, effectiveness, and safety of osteopathic manipulative treatment (OMT) using data collected from patients receiving OMT in the clinical setting within the established practice-based research network DO-Touch.NET.

. The HYPOTHESES of this research study are the following:

* OMT is primarily used in the treatment of musculoskeletal pain disorders.
* Patients receiving OMT will have decreased symptoms and improved quality-of-life.
* The most common side effect reported by patients receiving OMT will be muscle soreness.

DETAILED DESCRIPTION:
While many physicians and patients are convinced of the efficacy of osteopathic manipulative treatment (OMT), strong evidence supporting such a claim is sparse.

The objectives of this study are to determine the scope of conditions currently being treated with OMT, identify conditions that are responsive and unresponsive to OMT, determine which osteopathic manipulative techniques are most beneficial in responsive conditions, determine if certain patient characteristics are present in those who are responsive to OMT, and determine which physicians have consistently positive outcomes with OMT for certain conditions.

As an observational study, this study will not impact any aspect of the care received by the patient participants. Data will be collected from patients and physicians through a series of questionnaires incorporated into an online data collection system. DO-Touch.NET will be utilized for physician recruitment, site personnel training, members portal for accessing study materials, coordination, and physician data collection. Assessment Center will be used for participant registration, data collection and study tracking/reporting. Patients aged 18 years and older who receive OMT from a participating physician at a DO-Touch.NET site will be recruited to participate in the study. Background data will be collected from the patients including demographics, presenting symptoms and severity, and impact on quality of life. Data on medical history, examination, diagnosis, treatment, and home instructions/plan will be gathered from the physician. On a daily basis for a week after OMT, data will be collected from the patient regarding symptom severity and health changes. Impact of symptoms on quality of life will be reassessed after one week. These data will be collected from a patient over a series of office visits when applicable.

Ongoing observation of both positive and negative outcomes associated with OMT directly from patients will be increasingly more valuable, producing and sustaining a current evidence base for OMT and identifying priorities for further osteopathic research.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged 18 years and older
* Patients receiving OMT at a participating clinic

Exclusion Criteria:

* Patients with difficulty communicating in English, have dementia, or have psychological conditions that may impact their ability to provide accurate information
* Research team members and participating clinic employees

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study participants are recruited from participating physicians' office during patient hours for patients expected to receive OMT.
Sampling Method: Non-Probability Sample
Enrollment: 1960 (Actual)
Dates: Start 2011-07; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Pattern of Change in Severity of Chief Complaint | Baseline and 7 days following office visit
  Patient-reported severity level of chief complaint measured at baseline and daily for 7 days following office visit on an 11-point numeric rating scale (0=no problem, 10=worst imaginable).
Change in PROMIS Quality of Life Scales | Baseline to 1 week following office visit
  Select quality of life scales (fatigue, pain-interference, physical function, sleep disturbance) from the Patient Reported Outcomes Measurement Information System (PROMIS).
Patient-reported Assessment of Change in Overall Health Status | Immediately following office visit
  Assessment of how patient feels immediate following office visit overall compared to before office visit on 5-point ordinal scale (much better, better, about the same, worse, much worse)

CONTACTS AND LOCATIONS:
Overall Officials: Brian F Degenhardt, DO, Principal Investigator — A.T. Still Research Institute, A.T. Still University
Locations (17):
- United States (17):
  - Midwestern University Multispecialty Clinic, PC, Glendale, Arizona
  - Elizabeth M. Sasaki, DO, Visalia, California
  - Osteopathic Center for the Four Corners, Durango, Colorado
  - Rocky Mountain Integrative Medicine, Ridgway, Colorado
  - Feely Center of Optimal Health, Chicago, Illinois
  - Jefferson Park Medical Group, Chicago, Illinois
  - Midwestern University, Downers Grove, Illinois
  - Kohn Medical Group, McHenry, Illinois
  - New Medical Health Care, Wichita, Kansas
  - BMS Integrated Health, PLC, Farmington Hills, Michigan
  - Capital Region Medical Center, Jefferson City, Missouri
  - William James Brooks, DO, PC, Kansas City, Missouri
  - ATSU-KCOM OMM Clinic, Kirksville, Missouri
  - Kirksville Family Medicine, Kirksville, Missouri
  - Crossroads Premiere Health Care, Corvallis, Oregon
  - Walker Family Medicine, Winchester, Tennessee
  - Bee Caves Family Practice, Lakeway, Texas

REFERENCES:
- [Derived] Johnson JC, Degenhardt BF. Who Uses Osteopathic Manipulative Treatment? A Prospective, Observational Study Conducted by DO-Touch.NET. J Am Osteopath Assoc. 2019 Dec 1;119(12):802-812. doi: 10.7556/jaoa.2019.133. PMID 31790126
- See also: Practice based research network website. — http://www.DO-Touch.NET